CLINICAL TRIAL: NCT06370741
Title: Investigation of the Effectiveness of Achilles and Plantar Fascia-specific Stretching Methods on Plantar Fascia Mechanical Properties in Healthy Subjects: A Pilot Study
Brief Title: Effect of Stretching Exercises on Plantar Fascia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Ozgur Surenkok, Assistant professor, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: OkanUni.
Record Dates: First submitted 2024-04-05; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Stretch; Plantar Fascia; Contracture; Fasciitis, Plantar
MeSH Terms: conditions — Contracture; Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: Pilot study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Achilles tendon stretching (Experimental): Participants in this group will use a stretching device designed to stretch the dominant side Achilles tendon. With the help of this tool, the fingers will be positioned in extension and the other leg will be placed in front with the dominant side leg at the back. The knee of the other leg will be bent forward while the back knee is kept straight with the heel firmly on the ground. The toes of the evaluated foot will point to the heel of the front foot. For the non-dominant side, the same stretching exercise will be performed without equipment.
  Interventions: Device: Stretching with/without device
- Plantar fascia specific stretching (Active Comparator): A special stretching protocol known as PFSS (Plantar Fascia-Specific Stretching) will be applied. The method will be performed by placing the non-dominant leg over the opposite leg in a seated position. Following this, participants will apply force distal to the metatarsophalangeal joints in the assessed foot and pull the toes upwards towards the proximal side until a visible stretch is felt in the plantar fascia. Participants in this group will use the stretching device designed for their dominant side. The method will be performed by placing the toes on the bar of the device in the extension position and moving the knee forward so that the foot is in the dorsiflexion position without lifting the heel off the ground.
  Interventions: Device: Stretching with/without device

INTERVENTIONS:
Device: Stretching with/without device — Participants will be divided into two groups: Achilles tendon stretching and plantar fascia specific stretching. Within these two groups, participants will stretch their dominant side with the help of the designed tool. On the non-dominant side, the Achilles tendon group will complete the Achilles tendon stretching without a tool and the plantar fascia-specific stretching group will complete the self plantar fascia stretching exercise. Each stretching exercise will be performed for 10 seconds and 10 repetitions 3 days a week for 2 weeks.

SUMMARY:
The plantar fascia (PF) extends over the calcaneal bone with a thin band corresponding to the calcaneal periosteum, continuing as the paratenon of the Achilles tendon.The triceps surae complex, serving as the main extensor and propulsion system of the foot, involves the Achilles tendon, posterior part of the calcaneus, and Plantar Aponeurosis, all integrated with the fibrous skeleton of the triceps surae. Plantar fasciitis, a prevalent musculoskeletal condition affecting individuals of various ages and activity levels (Hye Chang Rhim), is a primary cause of heel pain in adults. Studies have identified the superior efficacy of stretching protocols targeting the Achilles tendon and/or plantar fascia compared to alternative treatments. However, the limitations of traditional approaches become apparent when considering the intricate biomechanics of the foot and ankle. Conventional calf stretches often prove inadequate for addressing its specific lengthening requirements. While contemporary methods like PF-Specific Stretching integrate plantar fascia and calf stretches, their reliance on individual upper extremity strength introduces potential limitations.

Therefore, although the exact effect of stretching on the biomechanical properties of the plantar fascia is not known, it will be aimed to determine whether an instrument aid to be designed will have an effect and which method is more effective. In this way, it is planned to guide clinicians in the rehabilitation of possible pathologies specific to the plantar fascia in clinical practice.

Myotonometry is a convenient method to assess the stiffness of the plantar fascia because it is cheap, simple and fast. Previous studies have shown that MyotonPRO can reliably assess the stiffness of the plantar fascia. Although the exact effect of stretching on the biomechanical properties of the plantar fascia is not known, it will be determined whether stretching with an instrument to be designed will have an effect and which method is more effective with or without an instrument.

DETAILED DESCRIPTION:
The intricate network of connective tissues in the foot, including the plantar aponeurosis (PA) originating from the calcaneus, sets the stage for a comprehensive understanding of conditions like plantar fasciitis. This broad and thick band runs longitudinally, forming distinct components crucial for maintaining the arch's integrity. Complementing this structure is the plantar fascia (PF), intricately connected to the superficial and deep muscles of the sole, creating a myofascial continuum with profound implications for foot biomechanics.

The interplay between the plantar fascia, Achilles tendon, and the Plantar Aponeurosis within the triceps surae complex emphasizes their collective role as the main extensor and propulsion system of the foot. The posterior compartment of the lower leg, housing various muscles, further underscores the complexity of this biomechanical system.

Nonoperative interventions, constituting approximately 90% effectiveness, encompass a range of approaches, including stretching exercises, modalities, and shock wave therapy, among others. Notably, studies have identified the superior efficacy of stretching protocols targeting the Achilles tendon and/or plantar fascia compared to alternative treatments.

However, the limitations of traditional approaches become apparent when considering the intricate biomechanics of the foot and ankle. Conventional calf stretches often prove inadequate for addressing its specific lengthening requirements. While contemporary methods like PF-Specific Stretching integrate plantar fascia and calf stretches, their reliance on individual upper extremity strength introduces potential limitations.

Myotonometry is a convenient method to assess the stiffness of the plantar fascia because it is cheap, simple and fast. Previous studies have shown that MyotonPRO can reliably assess the stiffness of the plantar fascia.

In the light of all this information, although the exact effect of stretching on the biomechanical properties of the plantar fascia is not known, it will be aimed to determine whether an instrument aid to be designed will have an effect and which method is more effective. In this way, it is planned to guide clinicians in the rehabilitation of possible pathologies specific to the plantar fascia in clinical practice.

Myotonometry is a convenient method to assess the stiffness of the plantar fascia because it is cheap, simple and fast. Previous studies have shown that MyotonPRO can reliably assess the stiffness of the plantar fascia. Although the exact effect of stretching on the biomechanical properties of the plantar fascia is not known, it will be determined whether stretching with an instrument to be designed will have an effect and which method is more effective with or without an instrument.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers over 18 years of age with a body mass index below 30 kg/m²

Exclusion Criteria:

* pregnancy, presence of chronic musculoskeletal diseases, presence of lower extremity injury and/or surgery, presence of skin lesions above the measurement sites and use of medications affecting the musculoskeletal system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Plantar Fascia Mechanical Properties | Before treatment/ Immediately after the first stretching exercise/ At the end of the second week
  MyotonPRO, an objective assessment method, will be used to evaluate the mechanical properties of the plantar fascia such as tone, stiffness and elasticity. MyotonPRO is a portable palpation device designed to assess the tone and biomechanical properties of muscle, tendon and fascia. This allows simultaneous calculation of the mechanical properties of the fascia: tonus - tension (frequency; Hz), stiffness - intramuscular resistance (N/m) and elasticity (characterized by decrement - logarithmic decrease)